CLINICAL TRIAL: NCT05983627
Title: A Clinical Trial to Evaluate the Safety, Tolerance and Efficacy of aCell Inj. of Allogeneic UC-MSCs in Patients With Mild to Moderate Acute Respiratory Distress Syndrome
Brief Title: Safety and Tolerance of Umbilical Cord Mesenchymal Stem Cells in Patients With Acute Respiratory Distress Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Asia Cell Therapeutics (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QS-ARDS-S1
Record Dates: First submitted 2023-07-26; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Human Umbilical Cord Mesenchymal Stem Cells; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord Mesenchymal Stem Cells (Experimental): The trial was divided into three dose groups： Low-dose group: 1000000 cells/kg Medium-dose group: 2000000 cells/kg High-does group: 4000000 cells/kg
  Interventions: Biological: Human Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Mesenchymal Stem Cells — The stem cell infusion route is peripheral intravenous infusion. All subjects received experimental drugs and conventional treatment during the study period.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of multiple doses of human umbilical cord mesenchymal stem cell injection in patients with Mild to Moderate Acute Respiratory Distress Syndrome (ARDS), and to further explore the efficacy, pharmacodynamic profile and appropriate dose of administration to provide a basis for the use of safer and more effective treatments for patients with Mild to Moderate Acute Respiratory Distress Syndrome (ARDS).

Participants are required to sign an informed consent form and, after undergoing a series of tests and meeting the protocol's entry and exclusion criteria, are assigned to a dose group for intravenous infusion of human umbilical cord mesenchymal stem cells. Each subject will receive three infusions.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) refers to various pathogenic factors that lead to excessive activation of the lung or even the whole body inflammatory response, which is manifested by the destruction of the lung epithelium and vascular endothelium, the decrease of alveolar clearance, and the occurrence of non-cardiogenic pulmonary edema. According to an international study involving 29144 patients, 10% of patients in ICU are ARDS patients, 23% of patients with mechanical ventilation suffer from ARDS, and the case fatality rate of ARDS ranges from 35% to 46%. At present, the treatment of ARDS includes primary disease treatment, protective mechanical ventilation and drug therapy, such as systemic infection, trauma, shock, burn, acute severe pancreatitis and other common causes of ARDS.

It is necessary to control the primary disease and control the systemic uncontrolled inflammatory response induced by it to prevent and treat ARDS. In the treatment of ARDS, in addition to actively treating the primary disease, respiratory support technology is the main treatment mode, which aims to correct intractable hypoxemia, prevent alveolar collapse, reduce the degree of pulmonary edema, improve the oxygenation index, and reduce respiratory muscle fatigue. In addition to the above treatment means, effective drug therapeutic intervention should be carried out early. Reducing ventilator dependence is the key to improve survival rate. Pharmacotherapy for ARDS includes anti-inflammatory drug therapy (such as glucocorticoids), antioxidant therapy for N-acetylcysteine, and alveolar surfactant replacement therapy.

Stem cells are a kind of undifferentiated cells that exist in embryonic or adult tissues and have the potential of self-renewal replication and multidirectional differentiation. mesenchymal stem cells (MSCs) are the most widely used stem cells in basic and clinical research. According to literature reports, MSCs have the ability to migrate to damaged tissues and repair damaged tissues through their multidirectional differentiation potential in vivo. Through its paracrine mechanism, MSCs can also improve the local microenvironment, support and promote the regeneration and differentiation of endogenous stem cells, play an anti-inflammatory role and regulate immunity. Human umbilical cord is considered medical waste and the collection of human umbilical cord mesenchymal stem cells is non-invasive, so there are no medical ethical issues with obtaining hUC-MSCs. Similar to other tissue-derived MSCs, hUC-MSCs have unique self-renewal ability and multi-differentiation potential, such as the ability to differentiate into adipose, bone, cartilage, nerve, and liver cells. Clinical trials of MSCs in the treatment of ARDS have been reported. A single-center, randomized, double-blind Phase I clinical trial reported the safety of intravenous injection of allogeneic adipose derived MSCs in the treatment of ARDS, and the results showed that MSCs were safe and non-tumorigenic. Another multi-center Phase I clinical trial reported the safety of different doses of MSCs derived from bone marrow in the treatment of ARDS. Based on this, the Phase II a clinical trial showed that MSCs improved the oxygenation index of ARDS patients. A case report reported that 2 patients with severe refractory ARDS showed improvement in respiratory distress, hemodynamic disturbance, and multiple organ failure after receiving MSCs treatment, which may be related to the reduction of inflammatory markers in the blood. The development of hUC-MSCs stem cell drugs has important clinical application value. At present, the human umbilical cord mesenchymal stem cell injection has completed the pharmacodynamics test of lung injury, the 4-week repeated administration in rats for 8 weeks, the 4-week repeated administration in rats for 8 weeks, the 4-week repeated administration in rhesus monkeys for 8 weeks, and the 4-week repeated administration in rhesus monkeys for 8 weeks Week recovery toxicity test, transfer and validation of toxic bioassay method (qPCR method), in vitro tumorigenesis test (soft AGAR cloning method), in vivo tumorigenesis test in naked mice (non-GLP), in vitro hemolysis test (rabbit blood), tissue distribution study in rats, safety pharmacological test of central nervous system in rats. In summary, the treatment of human umbilical cord mesenchymal stem cells has a wide safety window, and preclinical studies have shown that this product is safe and effective; The sponsors and investigators believe that MSC transplantation may improve the clinical symptoms of ARDS.

The clinical trial design of multi-center, single-arm, single administration, dose increment + dose extension was mainly adopted in this study. The "3+3" dose increment design was adopted in 3 preset dose groups, from low-dose group to high-dose group, and 3-6 subjects were included in each dose group Receive a corresponding dose. After all subjects in each dose group have completed the 2-week (14-day) DLT safety observation period, it will be up to the investigator and sponsor to discuss whether to proceed to the next dose group based on relevant safety data.

Adverse Events (AE) : All adverse medical events that occur after a clinical trial subject receives the investigational drug, but a clear causal relationship with the investigational drug may not be inferred. Adverse events can be symptoms, signs, diseases, or abnormalities in laboratory tests and include the following:

1. An aggravation of the pre-existing (prior to entry into the clinical trial) medical condition/disease (including an aggravation of symptoms, signs, laboratory abnormalities).
2. Any newly occurring adverse event: Any newly occurring adverse medical condition (including symptoms, signs, and newly diagnosed diseases).
3. Abnormal clinically significant laboratory test values or results that are not caused by concomitant disease.

Adverse reaction (ADR) : Any harmful or unintended reaction that may be associated with the investigational drug during a clinical trial. There is at least one reasonable possibility of a causal relationship between the investigational drug product and the adverse reaction, that is, an association cannot be ruled out.

Adverse events are monitored throughout the trial and it is the responsibility of the investigator to record all aes observed during the trial. The trial should record any adverse medical events, regardless of severity and causal relationship with the investigational drug, from the time of initial dosing until the end of follow-up, and the investigator should record them on the appropriate AE page in the CRF

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old (including the threshold), male or female
* A definite diagnosis of mild to moderate acute respiratory distress syndrome (ARDS) (according to the ARDS Berlin definition and diagnostic criteria)
* ARDS onset ≤ 5 days
* 100 mmHg < PaO2/FiO2 ≤ 300 mmHg
* Bilateral pulmonary infiltrates on chest radiograph or chest CT
* Rule out other causes of pulmonary oedema, such as cardiogenic pulmonary oedema and pulmonary oedema due to fluid overload
* Have no plans to have children within 2 weeks before screening and 3 months after the end of the trial, and agree to use effective non-pharmacological contraception during the trial
* Patients voluntarily signed an informed consent form and were willing to co-operate with the trial process

Exclusion Criteria:

* Hypersensitivity to known components of the drug (the main component of this product is human umbilical cord mesenchymal stem cells, excipients include dimethyl sulfoxide, human albumin, compound electrolyte injection), the presence of a history of allergy to gentamicin or other history of severe allergy
* Patients requiring treatment for any malignancy within 2 years prior to administration (except non-melanoma skin cancer)
* Lung transplant patients
* Patients with malignant haematological diseases
* Persons who have had a cardiovascular event within 3 months prior to dosing (e.g., unstable angina, congestive heart failure, myocardial infarction within the last 12 months, haemodynamic instability or known left ventricular ejection fraction (LVEF) <40% or clinically significant rhythm or conduction abnormalities)
* A history of deep vein thrombosis or pulmonary embolism during the Screening Period that, in the judgement of the Investigator, may be triggered or increase risk by receiving MSC transplantation therapy
* A breastfeeding female or a female with a positive blood pregnancy test result during the Screening Period
* History of immunodeficiency and/or autoimmune disease such as systemic lupus erythematosus (SLE), or other congenital immunodeficiency disease, idiopathic IgA deficiency. Laboratory tests at screening meet any of the following: Albuminous transaminase (AST) or albuminous transaminase (ALT) > 5 x ULN (non-hepatic sources are excluded; Serum creatinine > 1.5 x ULN or glomerular filtration rate < 60 mL/min/1.74 m2; Activated partial thromboplastin time (APTT) > 2.5 x ULN or prothrombin time; (PT) > 2.5 x ULN (not receiving anticoagulation)
* Positive infectious diseases (HBsAg, HCV, HIV-1, syphilis, active tuberculosis)
* Currently receiving extracorporeal life support (ECLS) such as continuous haemodialysis (CRRT) and carbon dioxide removal (ECCO2R), or high frequency oscillatory ventilation (HFOV)
* Presence of any other irreversible condition or symptom for which the subject has an expected survival of <3 months
* Combined WHO Class III or IV pulmonary hypertension
* Patients who refuse lung protective ventilation and fluid management
* Participation in other clinical trials or studies within 3 months prior to administration
* Persons with prior stem cell therapy
* Any other condition that, in the judgement of the investigator, makes participation in this trial inappropriate, such as a condition in which the study is not in the subject's current best interest (e.g., detrimental to health)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Day 1 to Day 28
  Adverse events that occurred during the trials
Serious Adverse Event (SAE) | Day 1 to Day 28
  Serious adverse events that occurred during the trial
Maximum Tolerated Dose (MTD) | Day 1 to Day 28
  Maximum Tolerated Dose

SECONDARY OUTCOMES:
Oxygenation index | Day 1(Before infusion)、Day 2、Day 3、Day 4、Day 7、Day 14、Day 28
  To observe the improvement in oxygenation index (P/F) from baseline
Chest routine scan | Baseline、Day 4、Day 14、Day 28
  To explore the improvement in lung imaging (calculation of lung exudate area)
Intubation rate | Day 1 to Day 28
  To explore the rate of intubation in subjects within 28 days after infusion
Length of hospitalisation | Day 1 to Day 28
  Length of stay in hospital within 28 days
Time out of ICU | Day 1 to Day 28
  Observe the time that subjects are not in the ICU for 28 days after infusion
Rate of Mortality | Day 1 to Day 28
  Rate of Mortality within 28 days after infusion
Murray lung injury score | Day 1(Before infusion)、Day 2、Day 3、Day 4、Day 7、Day 14、Day 28
  Improvement in assessment scores from baseline. The higher the score is, the more severe the lung damage is.

OTHER OUTCOMES:
Interferon-γ (IFN-γ） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、Day 28
  The concentration of IFN-γ in blood
Interleukin-1β （IL-1β） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、Day 28
  The concentration of IL-1β in blood
Interleukin-6 （IL-6） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、Day 28
  The concentration of IL-6 in blood
Interleukin-8 （IL-8） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、D28
  The concentration of IL-8 in blood
Interleukin-10 （IL-10） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、D28
  The concentration of IL-10 in blood
Tumor necrosis factor-α （TNF-α） | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、D28
  The concentration of TNF-α in blood
C-reaction protein (CRP) | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、D28
  The concentration of CRP in blood
Procalcitonin (PCT) | Baseline (1h before infusion)、Day 2、Day 3、Day 7、Day 14、Day 28
  The concentration of PCT in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, Principal Investigator — SHANGHAI JIAOTONG UNIVERSITY SCHOOL OF MEDICINE RUIJIN HOSPITAL